CLINICAL TRIAL: NCT00485589
Title: A Randomized, Double-Blind, Parallel Group, International Study to Evaluate the Safety and Efficacy of Ocrelizumab in Combination With Methotrexate (MTX) Compared to MTX Alone in Methotrexate- Naive Patients With Active Rheumatoid Arthritis
Brief Title: A Study of Ocrelizumab in Combination With Methotrexate in Patients With Rheumatoid Arthritis Who Are Naive to Methotrexate (FILM)
Acronym: FILM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Based on analysis of results and consideration of available treatments, the overall benefit to risk profile of ocrelizumab was not favorable in RA.
Sponsor: Genentech, Inc. (Industry)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACT3984g; WA20497
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Results first posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Rheumatoid Arthritis
Keywords: FILM; RA; anti-CD20; CD20
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; ocrelizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo (Placebo Comparator): Participants received placebo intravenously on Days 1 and 15 and Weeks 24, 26, 52, 54, 76, and 78. Participants also received methotrexate 7.5 mg orally weekly starting on Day 1. The dose of methodrexate was increased to a dose of 20 mg per week by Week 8, administered in 1 dose or divided into 3 equal doses administered at 12-hour intervals. Participants also received folate ≥ 5 mg/week either as a single dose or as a divided weekly dose. Participants were also allowed to continue receiving background corticosteroid therapy, at a dose of ≤ 10 mg/day of prednisolone or prednisolone.
  Interventions: Drug: Placebo
- Ocrelizumab 200 mg (Experimental): Participants received ocrelizumab 200 mg intravenously on Days 1 and 15 and Weeks 24, 26, 52, 54 and 76. Participants also received methotrexate 7.5 mg orally weekly starting on Day 1. The dose of methodrexate was increased to a dose of 20 mg per week by Week 8, administered in 1 dose or divided into 3 equal doses administered at 12-hour intervals. Participants also received folate ≥ 5 mg/week either as a single dose or as a divided weekly dose. Participants were also allowed to continue receiving background corticosteroid therapy, at a dose of ≤ 10 mg/day of prednisolone or prednisolone.
  Interventions: Drug: Methotrexate; Drug: Ocrelizumab
- Ocrelizumab 500 mg (Experimental): Participants received ocrelizumab 500 mg intravenously on Days 1 and 15 and Weeks 24, 26, 52, 54, and 76. Participants also received methotrexate 7.5 mg orally weekly starting on Day 1. The dose of methodrexate was increased to a dose of 20 mg per week by Week 8, administered in 1 dose or divided into 3 equal doses administered at 12-hour intervals. Participants also received folate ≥ 5 mg/week either as a single dose or as a divided weekly dose. Participants were also allowed to continue receiving background corticosteroid therapy, at a dose of ≤ 10 mg/day of prednisolone or prednisolone.
  Interventions: Drug: Methotrexate; Drug: Ocrelizumab

INTERVENTIONS:
Drug: Methotrexate — Oral repeating dose
  Arms: Ocrelizumab 200 mg; Ocrelizumab 500 mg
Drug: Ocrelizumab — Intravenous repeating dose
  Arms: Ocrelizumab 200 mg; Ocrelizumab 500 mg
Drug: Placebo — Intravenous repeating dose
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of ocrelizumab, compared with placebo, in combination with methotrexate in patients with active rheumatoid arthritis who are naive to methotrexate. Patients will be randomized to receive placebo, ocrelizumab 200mg i.v. or ocrelizumab 500mg i.v. on Days 1 and 15. Repeat courses of i.v. treatment will be administered at weeks 24, 52 and 76. All patients will receive concomitant methotrexate (7.5 mg escalating to 20mg p.o. weekly). The anticipated time on study treatment is 2+ years, and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18
* Rheumatoid arthritis for 3 months-5 years
* Naive to methotrexate
* If receiving steroids or NSAIDs, must be on a stable dose for 4 weeks prior to baseline

Exclusion criteria:

* Rheumatic autoimmune disease or inflammatory joint disease other than RA
* Prior receipt of any biologic therapy for RA
* Concurrent treatment with any DMARD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 613 (Actual)
Dates: Start 2007-06-11 (Actual); Primary Completion 2010-01-29 (Actual); Study Completion 2013-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Dummer, M.D., Study Director — Genentech, Inc.

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/members/ourmembers/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Emery P, Rigby W, Tak PP, Dorner T, Olech E, Martin C, Millar L, Travers H, Fisheleva E. Safety with ocrelizumab in rheumatoid arthritis: results from the ocrelizumab phase III program. PLoS One. 2014 Feb 3;9(2):e87379. doi: 10.1371/journal.pone.0087379. eCollection 2014. PMID 24498318

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study population comprised adult patients with active rheumatoid arthritis (RA) of at least 3 months' but less than 5 years' duration who were naïve to methotrexate. Additionally, patients were required to be naïve to any biologic therapy for RA prior to enrollment.
Period: Overall Study
Arm/Group | Placebo | Ocrelizumab 200 mg | Ocrelizumab 500 mg
Started | 210 | 200 | 203
Completed | 183 | 180 | 185
Not Completed | 27 | 20 | 18
Not completed — Death | 2 | 2 | 0
Not completed — Failure to return | 6 | 5 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Violation of selection criteria at entry | 0 | 3 | 1
Not completed — Administrative/Other | 1 | 2 | 1
Not completed — Insufficient therapeutic response | 10 | 3 | 1
Not completed — Refused treatment/did not cooperate | 1 | 0 | 2
Not completed — Withdrawal by Subject | 3 | 2 | 2
Not completed — Adverse Event | 3 | 3 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ocrelizumab 200 mg | Ocrelizumab 500 mg | Total
Number analyzed (Participants) | 207 | 196 | 202 | 605
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.2 (12.43) | 50.8 (13.17) | 48.6 (12.29) | 49.5 (12.66)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 153 | 154 | 161 | 468
  Male | 54 | 42 | 41 | 137

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Modified Total Sharp Score (mTSS) at Week 52
Description: The mTSS is a measure of joint damage and includes measures of joint erosion (JE) and joint space narrowing (JSN). The JE score, using the van der Heijde modification, measures erosion severity in 32 hand joints and 12 foot joints. Each hand joint is scored from 0 to 5 and each foot joint is scored from 0 to 10; the total score ranges from 0 to 280. Each joint is scored according to the surface area involved. A score of 10 indicates extensive loss of bone from more than one-half of the articulating bone; a score of 0 indicates no erosion. The JSN score measures the severity of JSN in 30 hand joints (15 per hand) and 12 foot joints (6 per foot). Each joint is scored from 0 to 4; the total score ranges from 0 to 168. A higher score indicates more joint space narrowing. The mTSS ranges from 0 to 448 (280+168). A higher mTSS score indicates greater damage. A negative change score indicates improvement.
Time Frame: Baseline to Week 52
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ocrelizumab 200 mg | Ocrelizumab 500 mg
Number analyzed (Participants) | 193 | 187 | 194
Units on a scale | 1.59 (4.815) | 0.66 (4.509) | 0.27 (2.908)
Statistical Analysis 1: Comparison: Placebo vs Ocrelizumab 200 mg; Test type: Non-Inferiority — Pre-specified analysis; p = 0.001, Van Elteren's test
Statistical Analysis 2: Comparison: Placebo vs Ocrelizumab 500 mg; Test type: Non-Inferiority — Pre-specified analysis; p = 0.0033, Van Elteren's test

2. Secondary Outcome: Percentage of Participants Without Radiographic Progression (RP) at Week 52
Description: RP was defined as a change from Baseline in the modified Total Sharp Score (mTSS) ≤ 0. The mTSS is a measure of joint damage and includes measures of joint erosion (JE) and joint space narrowing (JSN). The JE score, using the van der Heijde modification, measures erosion severity in 32 hand joints and 12 foot joints. Each hand joint is scored from 0 to 5 and each foot joint is scored from 0 to 10; the total score ranges from 0 to 280. Each joint is scored according to the surface area involved. A score of 10 indicates extensive loss of bone from more than one-half of the articulating bone; a score of 0 indicates no erosion. The JSN score measures the severity of JSN in 30 hand joints (15 per hand) and 12 foot joints (6 per foot). Each joint is scored from 0 to 4; the total score ranges from 0 to 168. A higher score indicates more joint space narrowing. The mTSS ranges from 0 to 448 (280+168). A higher mTSS score indicates greater damage. A negative change score indicates improvement.
Time Frame: Week 52
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Ocrelizumab 200 mg | Ocrelizumab 500 mg
Number analyzed (Participants) | 196 | 187 | 192
Percentage of participants | 51 [44 to 58] | 66.3 [59.5 to 73.1] | 68.8 [62.2 to 75.3]

3. Secondary Outcome: Percentage of Participants With an Improvement ≥ 20%, 50%, or 70% in American College of Rheumatology (ACR) Score (ACR20/50/70) From Baseline to Week 52
Description: Improvement must be seen in tender (68) and swollen (66) joint counts. Joints were assessed and classified as swollen/not swollen and tender/not tender by pressure and joint manipulation. Improvement must also be seen in at least 3 of the following 5 parameters: Separate patient and physician assessments of patient disease activity in the previous 24 hours on a visual analog scale (VAS, the extreme left end of the line "none" [symptom-free and no arthritis symptoms] and the extreme right end "maximum" [maximum arthritis disease activity]; patient assessment of pain in the previous 24 hours on a VAS (extreme left end of the line "none" and the extreme right end "unbearable"); Health Assessment Questionnaire-Disability Index (20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities, 0=without difficulty to 3=unable to do); and C-reactive protein (CRP), or erythrocyte sedimentation rate if CRP was missing.
Time Frame: Baseline to Week 52
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Ocrelizumab 200 mg | Ocrelizumab 500 mg
Number analyzed (Participants) | 207 | 196 | 200
Percentage of participants
  ACR20 | 57.5 [50.8 to 64.2] | 73 [66.7 to 79.2] | 71 [64.7 to 77.3]
  ACR50 | 39.6 [33 to 46.3] | 60.7 [53.9 to 67.6] | 54.5 [47.6 to 61.4]
  ACR70 | 20.3 [14.8 to 25.8] | 38.3 [31.5 to 45.1] | 38 [31.3 to 44.7]

4. Secondary Outcome: Percentage of Participants in Disease Activity Score 28 (DAS28) Remission at Weeks 24 and 52
Description: A participant was in DAS28 remission if their DAS28 score < 2.6). The DAS28 is a combined index for measuring disease activity in rheumatic arthritis (RA) and includes swollen and tender joint counts, erythrocyte sedimentation rate (ESR), and general health (GH) status. The index is calculated with the following formula: DAS28 = (0.56 × √(TJC28)) + (0.28 × √(SJC28)) + (0.7 × log(ESR)) + (0.014 × GH), where TJC28 = tender joint count and SJC28 = swollen joint count, each on 28 joints. GH = a patient's global assessment of disease activity in the previous 24 hours on a 100 mm visual analog scale (left end = no disease activity [symptom-free and no arthritis symptoms], right end = maximum disease activity [maximum arthritis disease activity]). When ESR equaled 0 mm/hr, it was set to 1 mm/hr. The DAS28 scale ranges from 0 to 10, where a higher score indicates more disease activity.
Time Frame: Week 24 and Week 52
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Ocrelizumab 200 mg | Ocrelizumab 500 mg
Number analyzed (Participants) | 207 | 196 | 200
Percentage of participants
  Week 24 | 9.7 [5.6 to 13.7] | 19.9 [14.3 to 25.5] | 18 [12.7 to 23.3]
  Week 52 | 7.2 [3.7 to 10.8] | 27 [20.8 to 33.3] | 28 [21.8 to 34.2]

ADVERSE EVENTS:
Time Frame: Baseline up to 30 months.
Description: Safety population: All randomized participants who received at least 1 dose of study medication.
Groups:
- Placebo - Treatment Period: Participants received placebo intravenously on Days 1 and 15 and Weeks 24, 26, 52, 54, 76 and 78. Participants also received methotrexate 20 mg orally per week by Week 8, administered in 1 dose or divided into 3 equal doses administered at 12-hour intervals. Participants also received acetaminophen 1 g and an antihistamine (diphenhydramine HCl 50 mg or equivalent dose of an alternative) orally 30-60 minutes prior to each infusion of study treatment and methylprednisolone 100 mg intravenously 30 minutes prior to each infusion of study treatment. Participants also received folate ≥ 5 mg/week either as a single dose or as a divided weekly dose. Participants were also allowed to continue receiving background corticosteroid therapy, at a dose of ≤ 10 mg/day of prednisolone.
- Placebo/Ocrelizumab 500 mg - Treatment Period: Participants received placebo intravenously on Days 1 and 15 and Weeks 24, 26, 52, 54, 76, and 78 and ocrelizumab 500 mg intravenously on Weeks 100, 102, 124, and 126. Participants also received methotrexate 20 mg orally per week by Week 8, administered in 1 dose or divided into 3 equal doses administered at 12-hour intervals. Participants also received acetaminophen 1 g and an antihistamine (diphenhydramine HCl 50 mg or equivalent dose of an alternative) orally 30-60 minutes prior to each infusion of study treatment and methylprednisolone 100 mg intravenously 30 minutes prior to each infusion of study treatment. Participants also received folate ≥ 5 mg/week either as a single dose or as a divided weekly dose. Participants were also allowed to continue receiving background corticosteroid therapy, at a dose of ≤ 10 mg/day of prednisolone.
- Ocrelizumab 200 mg - Treatment Period: Participants received placebo intravenously on Days 1 and 15 and Weeks 24, 26, 52, 54 and 76. Participants also received methotrexate 20 mg orally per week by Week 8, administered in 1 dose or divided into 3 equal doses administered at 12-hour intervals. Participants also received acetaminophen 1 g and an antihistamine (diphenhydramine HCl 50 mg or equivalent dose of an alternative) orally 30-60 minutes prior to each infusion of study treatment and methylprednisolone 100 mg intravenously 30 minutes prior to each infusion of study treatment. Participants also received folate ≥ 5 mg/week either as a single dose or as a divided weekly dose. Participants were also allowed to continue receiving background corticosteroid therapy, at a dose of ≤ 10 mg/day of prednisolone.
- Ocrelizumab 200 mg/Ocrelizumab 500 mg - Treatment Period: Participants received ocrelizumab 200 mg intravenously on Days 1 and 15 and Weeks 24, 26, 52, 54 and 76 and ocrelizumab 500 mg intravenously on Weeks 100, 102, 124, and 126. Participants also received methotrexate 20 mg orally per week by Week 8, administered in 1 dose or divided into 3 equal doses administered at 12-hour intervals. Participants also received acetaminophen 1 g and an antihistamine (diphenhydramine HCl 50 mg or equivalent dose of an alternative) orally 30-60 minutes prior to each infusion of study treatment and methylprednisolone 100 mg intravenously 30 minutes prior to each infusion of study treatment. Participants also received folate ≥ 5 mg/week either as a single dose or as a divided weekly dose. Participants were also allowed to continue receiving background corticosteroid therapy, at a dose of ≤ 10 mg/day of prednisolone.
- Ocrelizumab 500 mg - Treatment Period: Participants received ocrelizumab 500 mg intravenously on Days 1 and 15 and Weeks 24, 26, 52, 54 and 76. Participants also received methotrexate 20 mg orally per week by Week 8, administered in 1 dose or divided into 3 equal doses administered at 12-hour intervals. Participants also received acetaminophen 1 g and an antihistamine (diphenhydramine HCl 50 mg or equivalent dose of an alternative) orally 30-60 minutes prior to each infusion of study treatment and methylprednisolone 100 mg intravenously 30 minutes prior to each infusion of study treatment. Participants also received folate ≥ 5 mg/week either as a single dose or as a divided weekly dose. Participants were also allowed to continue receiving background corticosteroid therapy, at a dose of ≤ 10 mg/day of prednisolone.
- Ocrelizumab 500 mg/Ocrelizumab 500 mg - Treatment Period: Participants received ocrelizumab 500 mg intravenously on Days 1 and 15 and Weeks 24, 26, 52, 54, 76, 100, 102, 124, and 126. Participants also received methotrexate 20 mg orally per week by Week 8, administered in 1 dose or divided into 3 equal doses administered at 12-hour intervals. Participants also received acetaminophen 1 g and an antihistamine (diphenhydramine HCl 50 mg or equivalent dose of an alternative) orally 30-60 minutes prior to each infusion of study treatment and methylprednisolone 100 mg intravenously 30 minutes prior to each infusion of study treatment. Participants also received folate ≥ 5 mg/week either as a single dose or as a divided weekly dose. Participants were also allowed to continue receiving background corticosteroid therapy, at a dose of ≤ 10 mg/day of prednisolone.
- Placebo - Safety Follow-up Period: Participants had received placebo intravenously on Days 1 and 15 and Weeks 24, 26, 52, 54, 76 and 78. Participants also received methotrexate 20 mg orally per week by Week 8, administered in 1 dose or divided into 3 equal doses administered at 12-hour intervals. Participants also received acetaminophen 1 g and an antihistamine (diphenhydramine HCl 50 mg or equivalent dose of an alternative) orally 30-60 minutes prior to each infusion of study treatment and methylprednisolone 100 mg intravenously 30 minutes prior to each infusion of study treatment. Participants also received folate ≥ 5 mg/week either as a single dose or as a divided weekly dose. Participants were also allowed to continue receiving background corticosteroid therapy, at a dose of ≤ 10 mg/day of prednisolone.
- Placebo/Ocrelizumab 500 mg - Safety Follow-up Period: Participants had received placebo intravenously on Days 1 and 15 and Weeks 24, 26, 52, 54, 76, and 78 and ocrelizumab 500 mg intravenously on Weeks 100, 102, 124, and 126. Participants also received methotrexate 20 mg orally per week by Week 8, administered in 1 dose or divided into 3 equal doses administered at 12-hour intervals. Participants also received acetaminophen 1 g and an antihistamine (diphenhydramine HCl 50 mg or equivalent dose of an alternative) orally 30-60 minutes prior to each infusion of study treatment and methylprednisolone 100 mg intravenously 30 minutes prior to each infusion of study treatment. Participants also received folate ≥ 5 mg/week either as a single dose or as a divided weekly dose. Participants were also allowed to continue receiving background corticosteroid therapy, at a dose of ≤ 10 mg/day of prednisolone.
- Ocrelizumab 200 mg - Safety Follow-up Period: Participants had received Ocrelizumab intravenously on Days 1 and 15 and Weeks 24, 26, 52, 54 and 76. Participants received methotrexate 20 mg orally per week by Week 8, administered in 1 dose or divided into 3 equal doses administered at 12-hour intervals. Participants also received acetaminophen 1 g and an antihistamine (diphenhydramine HCl 50 mg or equivalent dose of an alternative) orally 30-60 minutes prior to each infusion of study treatment and methylprednisolone 100 mg intravenously 30 minutes prior to each infusion of study treatment. Participants also received folate ≥ 5 mg/week either as a single dose or as a divided weekly dose. Participants were also allowed to continue receiving background corticosteroid therapy, at a dose of ≤ 10 mg/day of prednisolone.
- Ocrelizumab 200 mg/Ocrelizumab 500 Mg-safety Follow-up Period: Participants had received ocrelizumab 200 mg intravenously on Days 1 and 15 and Weeks 24, 26, 52, 54 and 76 and ocrelizumab 500 mg intravenously on Weeks 100, 102, 124, and 126. Participants also received methotrexate 20 mg orally per week by Week 8, administered in 1 dose or divided into 3 equal doses administered at 12-hour intervals. Participants also received acetaminophen 1 g and an antihistamine (diphenhydramine HCl 50 mg or equivalent dose of an alternative) orally 30-60 minutes prior to each infusion of study treatment and methylprednisolone 100 mg intravenously 30 minutes prior to each infusion of study treatment. Participants also received folate ≥ 5 mg/week either as a single dose or as a divided weekly dose. Participants were also allowed to continue receiving background corticosteroid therapy, at a dose of ≤ 10 mg/day of prednisolone.
- Ocrelizumab 500 mg - Safety Follow-up Period: Participants had received ocrelizumab 500 mg intravenously on Days 1 and 15 and Weeks 24, 26, 52, 54, 76 and 78. Participants also received methotrexate 20 mg orally per week by Week 8, administered in 1 dose or divided into 3 equal doses administered at 12-hour intervals. Participants also received acetaminophen 1 g and an antihistamine (diphenhydramine HCl 50 mg or equivalent dose of an alternative) orally 30-60 minutes prior to each infusion of study treatment and methylprednisolone 100 mg intravenously 30 minutes prior to each infusion of study treatment. Participants also received folate ≥ 5 mg/week either as a single dose or as a divided weekly dose. Participants were also allowed to continue receiving background corticosteroid therapy, at a dose of ≤ 10 mg/day of prednisolone.
- Ocrelizumab 500 mg/Ocrelizumab 500 mg -Safety Follow-up Period: Participants had received ocrelizumab 500 mg intravenously on Days 1 and 15 and Weeks 24, 26, 52, 54, 76, 100, 102, 124, and 126. Participants also received methotrexate 20 mg orally per week by Week 8, administered in 1 dose or divided into 3 equal doses administered at 12-hour intervals. Participants also received acetaminophen 1 g and an antihistamine (diphenhydramine HCl 50 mg or equivalent dose of an alternative) orally 30-60 minutes prior to each infusion of study treatment and methylprednisolone 100 mg intravenously 30 minutes prior to each infusion of study treatment. Participants also received folate ≥ 5 mg/week either as a single dose or as a divided weekly dose. Participants were also allowed to continue receiving background corticosteroid therapy, at a dose of ≤ 10 mg/day of prednisolone.
Arm/Group | Placebo - Treatment Period | Placebo/Ocrelizumab 500 mg - Treatment Period | Ocrelizumab 200 mg - Treatment Period | Ocrelizumab 200 mg/Ocrelizumab 500 mg - Treatment Period | Ocrelizumab 500 mg - Treatment Period | Ocrelizumab 500 mg/Ocrelizumab 500 mg - Treatment Period | Placebo - Safety Follow-up Period | Placebo/Ocrelizumab 500 mg - Safety Follow-up Period | Ocrelizumab 200 mg - Safety Follow-up Period | Ocrelizumab 200 mg/Ocrelizumab 500 Mg-safety Follow-up Period | Ocrelizumab 500 mg - Safety Follow-up Period | Ocrelizumab 500 mg/Ocrelizumab 500 mg -Safety Follow-up Period
All-Cause Mortality (participants affected / at risk) | 0/207 | 0/10 | 0/196 | 0/12 | 0/202 | 0/6 | 2/187 | 0/9 | 2/177 | 0/11 | 1/185 | 0/6
Serious Adverse Events (participants affected / at risk) | 22/207 | 0/10 | 21/196 | 1/12 | 31/202 | 0/6 | 11/187 | 2/9 | 2/177 | 0/11 | 4/185 | 0/6
Other Adverse Events (participants affected / at risk) | 128/207 | 4/10 | 135/196 | 6/12 | 144/202 | 3/6 | 35/187 | 3/9 | 32/177 | 3/11 | 49/185 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Treatment Period (N=207) | Placebo/Ocrelizumab 500 mg - Treatment Period (N=10) | Ocrelizumab 200 mg - Treatment Period (N=196) | Ocrelizumab 200 mg/Ocrelizumab 500 mg - Treatment Period (N=12) | Ocrelizumab 500 mg - Treatment Period (N=202) | Ocrelizumab 500 mg/Ocrelizumab 500 mg - Treatment Period (N=6) | Placebo - Safety Follow-up Period (N=187) | Placebo/Ocrelizumab 500 mg - Safety Follow-up Period (N=9) | Ocrelizumab 200 mg - Safety Follow-up Period (N=177) | Ocrelizumab 200 mg/Ocrelizumab 500 Mg-safety Follow-up Period (N=11) | Ocrelizumab 500 mg - Safety Follow-up Period (N=185) | Ocrelizumab 500 mg/Ocrelizumab 500 mg -Safety Follow-up Period (N=6)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dislocation of vertebra (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchogenic cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary eosinophilia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Autonomic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness bilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal wall infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0
Encephalitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Histoplasmosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia herpes viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.05% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Treatment Period (N=207) | Placebo/Ocrelizumab 500 mg - Treatment Period (N=10) | Ocrelizumab 200 mg - Treatment Period (N=196) | Ocrelizumab 200 mg/Ocrelizumab 500 mg - Treatment Period (N=12) | Ocrelizumab 500 mg - Treatment Period (N=202) | Ocrelizumab 500 mg/Ocrelizumab 500 mg - Treatment Period (N=6) | Placebo - Safety Follow-up Period (N=187) | Placebo/Ocrelizumab 500 mg - Safety Follow-up Period (N=9) | Ocrelizumab 200 mg - Safety Follow-up Period (N=177) | Ocrelizumab 200 mg/Ocrelizumab 500 Mg-safety Follow-up Period (N=11) | Ocrelizumab 500 mg - Safety Follow-up Period (N=185) | Ocrelizumab 500 mg/Ocrelizumab 500 mg -Safety Follow-up Period (N=6)
Hypertension (Vascular disorders) | 23 (23) | 0 (0) | 14 (14) | 0 (0) | 18 (18) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bunion operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 21 (36) | 4 (4) | 56 (79) | 0 (0) | 64 (91) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (3) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Sinusitis noninfective (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 13 (13) | 0 (0) | 12 (12) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 24 (24) | 0 (0) | 16 (16) | 0 (0) | 22 (22) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 14 (14) | 0 (0) | 7 (7) | 0 (0) | 14 (14) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 14 (14) | 0 (0) | 8 (8) | 0 (0) | 13 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0) | 0 (0)
Gastritis atrophic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 18 (18) | 0 (0) | 28 (28) | 0 (0) | 27 (27) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 0 (0) | 10 (10) | 0 (0) | 7 (7) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 6 (7) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 36 (45) | 0 (0) | 31 (38) | 0 (0) | 23 (29) | 1 (1) | 7 (7) | 1 (1) | 3 (3) | 2 (3) | 7 (7) | 0 (0)
Cystitis (Infections and infestations) | 3 (4) | 0 (0) | 4 (6) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 21 (21) | 0 (0) | 22 (22) | 0 (0) | 15 (15) | 0 (0) | 3 (3) | 1 (1) | 5 (5) | 0 (0) | 3 (5) | 0 (0)
Urinary tract infection (Infections and infestations) | 12 (12) | 0 (0) | 21 (21) | 0 (0) | 25 (25) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 12 (12) | 0 (0)
Nasopharyngitis (Infections and infestations) | 11 (11) | 0 (0) | 18 (18) | 0 (0) | 16 (16) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 10 (10) | 0 (0) | 7 (7) | 0 (0) | 15 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 9 (9) | 0 (0) | 10 (10) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 3 (4) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated prematurely by the sponsors before all patients could reach the time point for primary analysis at Week 104. No patient received any further infusions of study medication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.